CLINICAL TRIAL: NCT03643861
Title: RAD 1802: A Pilot Trial of Five Fraction Stereotactic Body Radiotherapy for Early Stage Breast Cancer Patients Eligible for Post-Operative Accelerated Partial Breast Irradiation (APBI)
Brief Title: RAD 1802: Pilot Trial of Five Fraction Stereotactic Body Radiotherapy for Early Stage Breast Cancer Patients Eligible for Post-Operative Accelerated Partial Breast Irradiation (APBI)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Principal Investigator, Drexell Hunter Boggs, Radiation Oncologist, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300002157; 000521633 (Other Grant/Funding Number: Varian Medical Systems)
Record Dates: First submitted 2018-08-17; First posted 2018-08-23 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer
Keywords: SBRT; Breast cancer; Early stage; Radiation therapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- 5 Fraction Breast Stereotactic Body Radiation Therapy (Experimental): This study will enroll patients that have a confirmed histology of early stage breast cancer. The patient will undergo a lumpectomy and will then receive partial breast 5 fractions stereotactic body radiation therapy at a dose of 6 gy for 5 fractions for treatment. Patients will be followed for 36 total months with specific follow-ups at 3, 6, 9, 12, 18, 24, and 36 months.
  Interventions: Radiation: 5 Fraction Stereotactic Body Radiation Therapy

INTERVENTIONS:
Radiation: 5 Fraction Stereotactic Body Radiation Therapy — Stereotactic body radiation therapy (SBRT) has gained favor in the treatment of select central nervous system, lung, and abdominal malignancies due to its ability to deliver highly conformal doses of radiotherapy while using sharp dose gradients to deliver comparatively lower doses to the surrounding normal tissue. Utilization of SBRT is more labor intensive than conventional fractionation and requires precise immobilization and localization techniques with daily image guidance with direct physician and physicist oversight for all treatments. While more labor intensive and often utilizing more advanced technologies, SBRT allows the advantage of reducing setup margins compared to conventionally fractionated treatment while being able to shorten overall treatment times due to the ability to safely dose escalate high risk areas

SUMMARY:
This study offers 5 fractions of radiation treatment through partial breast irradiation in patients with early stage breast cancer after having a lumpectomy.

DETAILED DESCRIPTION:
This study offers 5 fractions stereotactic body radiotherapy for early stage breast cancer after patient undergoes a lumpectomy. The study aims to determine the safety and feasibility of delivering only 5 doses of radiation treatment rather than the longer schedule of treatments that is currently considered standard of care for breast cancer patients. Patients will be followed for 36 months (2 years) with follow-up appointments at 6, 12, 18, 24, and 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven invasive mammary carcinoma, Invasive ductal carcinoma (IDC) or ductal carcinoma in situ (DCIS) of the breast. Medullary, papillary, mucinous (colloid) and tubular histologies are allowed.
* Age>50.
* Maximum pathologic tumor size <2.0cm if invasive carcinoma or < 2.5cm if pure DCIS.
* Estrogen receptor (ER) positive (>10%).
* Must be eligible for breast conservation therapy and receive a lumpectomy with pathologic margins of at least 2mm.
* Must be clinically node negative by physical examination. Sentinel node dissection is not required, but if undertaken, the patient must be pathologically node negative.
* Zubrod Performance Status 0-2.

Exclusion Criteria:

* Multifocal or multicentric cancer.
* Reception of neoadjuvant chemotherapy.
* Pure invasive lobular histology.
* Inability to clearly delineate lumpectomy cavity on post lumpectomy planning scan.
* Measured maximum PTV of >124cc.
* Lumpectomy cavity within 5mm of body contour.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-08-20 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Toxicity levels of 5 fractions SBRT for partial breast irradiation assessed by CTCAE v4.0 | 0-2 years
  To determine the safety of 5 fractions SBRT for patients with early stage breast cancer after a lumpectomy. Safety will be determined by CTCAE v4.0 and access toxicity, or lack of, experienced by patients enrolled in this study.

SECONDARY OUTCOMES:
Toxicity of breast SBRT using CTCAE v4.0 | 0-2 years
  To define the acute (<90 days) and late toxicity (>90 days) up to two years after breast SBRT (CTCAE 4) attributable to therapy.
Cosmetic outcome baseline and post-SBRT | 0-2 years
  To determine patient and nurse assessed cosmetic outcome at baseline and 1, 6, 12, 18, 24, and 36 months post SBRT. Patient will give a verbal satisfaction rating of 1-Excellent, 2-Good, 3-Fair, or 4-Poor of their cosmetic appearance post-SBRT. Nurse will also give their overall rating of 1-Excellent, 2-Good, 3-Fair, or 4-Poor based off of their examination of the cosmetic appearance post-SBRT.
Patient reported outcome baseline and post-SBRT | 0-2 years
  To determine patient reported outcome at baseline and 1, 6, 12, 18, 24, and 36 months post SBRT. The Quality of Life Breast Cancer Questionnaire (QLQ-BR45) is a 45-item questionnaire is composed of 45 questions with scale of 4 options where 1 represents "not at all" to 4 "very much". Scores on the QLQ-BR45 range from 45 to 180, with a lower score representing a higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: D. Hunter Boggs, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham (UAB) Hazelrig-Salter Radiation Oncology Center (HSROC), Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liu Y, Veale C, Hablitz D, Krontiras H, Dalton A, Meyers K, Dobelbower M, Lancaster R, Bredel M, Parker C, Keene K, Thomas E, Boggs D. Feasibility and Short-Term Toxicity of a Consecutively Delivered Five Fraction Stereotactic Body Radiation Therapy Regimen in Early-Stage Breast Cancer Patients Receiving Partial Breast Irradiation. Front Oncol. 2022 Jul 8;12:901312. doi: 10.3389/fonc.2022.901312. eCollection 2022. PMID 35880164